CLINICAL TRIAL: NCT02682420
Title: everlinQ endoAVF Post Market Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company acquisition
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-0018
Record Dates: First submitted 2016-02-05; First posted 2016-02-15 (Estimated); Results first posted 2021-11-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endoAVF (Other)
  Interventions: Device: everlinQ endoAVF System

INTERVENTIONS:
Device: everlinQ endoAVF System

SUMMARY:
Prospective, multi-center study to evaluate the everlinQ endoAVF System when used to create an endovascular arteriovenous fistula (endoAVF) for patients who require vascular access for hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age >18 years old)
* Currently on chronic dialysis or expected to be started on chronic dialysis within 3 months of planned endoAVF creation
* Target treatment vein diameter(s) for fistula creation ≥ 2.0 mm as measured via Duplex Ultrasound or Venogram
* Target treatment artery diameter(s) for fistula creation ≥ 2.0 mm as measured via Duplex Ultrasound or Arteriogram
* Both radial and ulnar artery flow to the hand, as confirmed with Duplex Ultrasound and/or Allen's test (i.e.: palmar arch)

Exclusion Criteria:

* Known central venous stenosis or central vein narrowing > 50% based on imaging on the same side as the planned AVF creation
* Absence of perforator feeding the target cannulation vein(s) via Venogram
* Occlusion or stenosis >50% of target cannulation cephalic or basilic vein
* Significantly compromised (≥50% stenosis) flow in the treatment arm
* Documented ejection fraction (EF) ≤35% in the last 6 months
* Pregnant women
* New York Heart Association (NYHA) class III or IV heart failure
* Hypercoagulable state
* Known bleeding diathesis
* Documented history of drug abuse including intravenous drugs within six months of AVF creation
* "Planned" concomitant major surgical procedure within 6 months of enrollment or previous major surgery within 30 days of enrollment
* Known allergy to contrast dye which cannot be adequately pre-medicated
* Known adverse effects to sedation and/or anesthesia which cannot be adequately pre-medicated
* Evidence of active infections on the day of the index procedure
* Estimated life expectancy < 1 year
* Patient is not willing to provide written informed consent, is not geographically stable and/or not willing to comply with required follow-up
* Patient with a target cannulation vein that is > 6mm deep that would require a transposition procedure, defined as the elevation of a target cannulation vein AND the creation of a new AV fistula
* Patient is not willing to undergo a 2nd stage procedure as defined in Section 4.5.3 of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Inston, MD, Principal Investigator — University Hospitals Birmingham NHS; Thomas Schmitz-Rixen, MD, Principal Investigator — Univerisity of Frankfurt, Germany
Locations (11):
- Providence Health Care Society, Vancouver, British Columbia, Canada
- Germany (6):
  - University Hospital Carl Gustav Carus, Dresden
  - Dominikus Hospital, Düsseldorf
  - University of Frankfurt, Frankfurt
  - University of Leipzig, Leipzig
  - University of Mannheim, Mannheim
  - St. Franziskus-Hospital Münster, Münster
- United Kingdom (4):
  - Oxford University Hospitals - NHS Foundation Trust, Headington, Oxford
  - University Hospitals Birmingham, Birmingham
  - St. George's University, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The everlinQ endoAVF Post Market Study began enrollment on September 20th 2016 and the last patient was enrolled on January 17th 2019.
Groups:
- endoAVF: everlinQ endoAVF System: The everlinQ device is a single-use disposable device. The everlinQ catheter system consists of two flexible, magnetic catheters. Once the catheters are properly inserted and aligned, the magnets contained in each catheter attract to one another, approximating the vessels while simultaneously aligning the electrode with the backstop. Radiofrequency (RF) energy is delivered to the electrode whereby the arterio-venous fistula (AVF) is created.
Period: Overall Study
Arm/Group | endoAVF
Started | 100
Completed | 63 (Note: 63 participants completed the 6-month visit. The study was discontinued prematurely due to company acquisition and therefore, many participants did not complete their 12-month visit.)
Not Completed | 37

BASELINE CHARACTERISTICS:
Groups:
- endoAVF: everlinQ endoAVF System: The everlinQ device is a single-use disposable device. The everlinQ catheter system consists of two flexible, magnetic catheters. Once the catheters are properly inserted and aligned, the magnets contained in each catheter attract to one another, approximating the vessels while simultaneously aligning the electrode with the backstop. RF energy is delivered to the electrode whereby the arterio-venous fistula (AVF) is created.
Arm/Group | endoAVF
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 70
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  Canada | 14
  United Kingdom | 59
  Germany | 26
  Netherlands | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (7.6)
EndoAVF Device [Count of Participants; unit: Participants] — This baseline measure describes the everlinQ endoAVF device selected by the physician for the participant's index procedure. Two different size devices were used within this study: the 4 French version and the 6 French version.
  Participants
    4 French | 64
    6 French | 36

OUTCOME MEASURES:

1. Primary Outcome: Participants With Primary Patency of the endoAVF at 6 Months Post-Index Procedure
Description: Primary patency was defined in this study as "The interval from the time of access placement until any intervention designed to maintain or re-establish patency, access thrombosis, access abandonment, or the time of measurement of patency".
Time Frame: endoAVF creation through 6 months
Measure: Number; unit: percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 54
percentage of participants | 71

2. Other Pre Specified Outcome: Participants With Assisted Primary Patency of the endoAVF at 6 Months Post-Index Procedure
Description: Assisted Primary Patency was defined in this study as "The interval from access placement to thrombosis or abandonment; not triggered by access circuit interventions performed in the absence of occlusion".
Time Frame: endoAVF creation through 6 Months
Measure: Number; unit: percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 52
percentage of participants | 81

3. Other Pre Specified Outcome: Participants With Secondary Patency of the endoAVF at 6 Months Post-Index Procedure
Description: Secondary Patency in this study was defined as "The interval from the time of access placement until access abandonment, loss to thrombosis, or the time of patency measurement including intervening manipulations (surgical or endovascular interventions) designed to re-establish functionality in thrombosed access".
Time Frame: endoAVF creation through 6 Months
Measure: Number; unit: percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 62
percentage of participants | 91

4. Other Pre Specified Outcome: Participants With Functional Patency of the endoAVF at 6 Months Post-Index Procedure
Description: Functional Patency in this study was defined as "The interval of time from the first 2-needle dialysis utilizing the access until access abandonment".
Time Frame: endoAVF creation through 6 Months
Measure: Number; unit: percentage of participants
Arm/Group | endoAVF
Number analyzed (Participants) | 20
percentage of participants | 95

5. Other Pre Specified Outcome: Number of Days Post-Index Procedure for Participants to Achieve Successful Cannulation of the endoAVF
Description: The time (number of days) from the index procedure (successful endoAVF creation) to the first use of the endoAVF. This endpoint is evaluated per participant rather than at specific time points.
Time Frame: endoAVF creation to cannulation
Population: Only participants remaining in the study that were on dialysis can be counted for this endpoint.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | endoAVF
Number analyzed (Participants) | 50
days | 84 [60 to 139]

6. Other Pre Specified Outcome: Number of Participants With Procedural Success at the Index Procedure
Description: The successful creation of an endoAVF with blood flow confirmed intraoperatively by fistulography or by duplex ultrasound postoperatively. This outcome measure is assessed at the time of the endoAVF creation.
Time Frame: endoAVF creation
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 100
Participants | 94

7. Other Pre Specified Outcome: Number of Participants With Interventions Occurring During the Index Procedure (Adjunctive Procedures)
Description: The endoAVF-related interventions include:
  * Interventions to maintain or restore patency of the endoAVF, including endovascular and surgical procedures designed to address occlusive thrombosis (resulting in absence of thrill or bruit at endoAVF) and clinically significant occlusive stenosis at or near endoAVF site.
  * Interventions to support maturation of the arterialized vein segments, including endovascular procedures such as secondary coil embolization to facilitate flow into the target cannulation veins.
  * Interventions to support cannulation of the arterialized vein segments, including procedures such as a superficialization or elevation where the target cannulation vein is brought closer to the skin surface to enable cannulation, without the creation of a new AV fistula.
  * Any intervention to address any complications or adverse events of the access circuit.
  This outcome measure is assessed at the time of the endoAVF creation.
Time Frame: endoAVF creation
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 100
Participants
  Therapeutic Coil Embolization | 73
  Balloon Angioplasty | 0
  Stent | 0
  Thrombectomy | 0
  Thrombolytic Therapy | 0
  Transposition | 2
  Creation of Surgical AVF/Graft | 0
  Other | 0
  Participants with ≥1 Adjunctive Procedures | 74

8. Other Pre Specified Outcome: Number of Participants With Interventions Occurring After the Index Procedure (Reinterventions)
Description: The endoAVF-related interventions include:
  * Interventions to maintain or restore patency of the endoAVF, including endovascular and surgical procedures designed to address occlusive thrombosis (resulting in absence of thrill or bruit at endoAVF) and clinically significant occlusive stenosis at or near endoAVF site.
  * Interventions to support maturation of the arterialized vein segments, including endovascular procedures such as secondary coil embolization to facilitate flow into the target cannulation veins.
  * Interventions to support cannulation of the arterialized vein segments, including procedures such as a superficialization or elevation where the target cannulation vein is brought closer to the skin surface to enable cannulation, without the creation of a new AV fistula.
  * Any intervention to address any complications or adverse events of the access circuit.
Time Frame: endoAVF creation through 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 100
Participants
  Total Maturation and Maintenance Interventions | 26
  Subjects with ≥1 Reintervention | 24
  Total Maturation Interventions | 18
  Superficialization (Maturation) | 10
  Coiling (Maturation) | 8
  Total Maintenance Interventions | 8
  PTA (Maintenance) | 6
  Stent Placement (Maintenance) | 1
  Thrombolysis (Maintenance) | 1

9. Other Pre Specified Outcome: Participants in Which endoAVF Maturation Was Achieved
Description: Total time from successful endoAVF creation to one of the following:
  * Successful hemodialysis using 2 needle cannulation OR
  * Vascular access that is free of stenosis or thrombosis, with brachial artery flow of at least 500 ml/min and at least a 4.0 mm vein diameter as measured via duplex ultrasound.
  Note: 63 participants completed the 6-month visit. Participants who did not receive a duplex ultrasound and have not yet successfully dialyzed using 2 needle cannulation are not counted for this endpoint.
Time Frame: endoAVF creation through 6 months
Measure: Count of Participants; unit: Participants
Groups:
- At 1 Month: Participants that have met the definition for maturity by the 1 Month follow-up visit
- At 3 Months: Participants that have met the definition for maturity by the 3 Month follow-up visit
- At 6 Months: Participants that have met the definition for maturity by the 6 Month follow-up visit
- At Any Visit: Participants that have met the definition for maturity at any visit
Arm/Group | At 1 Month | At 3 Months | At 6 Months | At Any Visit
Number analyzed (Participants) | 79 | 70 | 57 | 91
Participants | 63 | 59 | 47 | 83

10. Other Pre Specified Outcome: Number of Participants That Were Not on Dialysis at endoAVF Creation and Are Central Venous Catheter (CVC) Free at Indicated Time Points
Description: Number of participants that were not on dialysis at endoAVF creation and are central venous catheter (CVC) free at indicated time points.
Time Frame: endoAVF creation through 6 Months
Measure: Count of Participants; unit: Participants
Groups:
- At 1 Month: Participants that were not on dialysis at the time of endoAVF creation and were catheter-free at 30 days of follow-up
- At 6 Months: Participants that were not on dialysis at the time of endoAVF creation and were catheter-free at 180 days of follow-up
Arm/Group | At 1 Month | At 6 Months
Number analyzed (Participants) | 24 | 24
Participants | 22 | 23

11. Other Pre Specified Outcome: Number of Participants That Experienced Device-related Serious Adverse Events Through 6 Months Post-Index Procedure
Description: AE that:
  * led to death,
  * led to serious deterioration in the health of the patient, that either resulted in: a life-threatening illness or injury, or a permanent impairment of a body structure or a body function, or in-patient or prolonged hospitalization, or medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
  * led to fetal distress, fetal death or a congenital abnormality or birth defect And has been determined by the CEC to be related to the everlinQ endoAVF System
Time Frame: endoAVF creation through 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 100
Participants | 3

12. Other Pre Specified Outcome: Number of Participants That Experienced Procedure-related Serious Adverse Events Through 6 Months Post-Index Procedure
Description: AE that:
  * led to death,
  * led to serious deterioration in the health of the patient, that either resulted in: a life-threatening illness or injury, or a permanent impairment of a body structure or a body function, or in-patient or prolonged hospitalization, or medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
  * led to fetal distress, fetal death or a congenital abnormality or birth defect And has been determined by the CEC to be related to the index procedure
Time Frame: endoAVF creation through 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | endoAVF
Number analyzed (Participants) | 100
Participants | 11

13. Post Hoc Outcome: Dialysis Status
Description: This outcome measure references the participant's dialysis status throughout the study. Participants who began dialysis during the study and participants who were not on dialysis through the end of the study were not on dialysis at baseline.
Time Frame: endoAVF creation through 6 months
Measure: Number; unit: participants
Arm/Group | endoAVF
Number analyzed (Participants) | 100
participants
  On Dialysis at Enrollment | 47
  Began Dialysis During Study | 24
  Not on Dialysis Through End of Study | 29

ADVERSE EVENTS:
Time Frame: Adverse events were reported from index procedure through the study follow-up period. Data is reported through 6 months.
Arm/Group | endoAVF
All-Cause Mortality (participants affected / at risk) | 3/100
Serious Adverse Events (participants affected / at risk) | 24/100
Other Adverse Events (participants affected / at risk) | 7/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | endoAVF (N=100)
Stenosis (Vascular disorders) | 5 (5)
Pseudoaneurysm (Vascular disorders) | 3 (3)
Bruising/Hematoma (Blood and lymphatic system disorders) | 3 (3)
Thrombosis (Vascular disorders) | 4 (4)
Compartment Syndrome (Blood and lymphatic system disorders) | 2 (2)
Closure Device Embolization (Blood and lymphatic system disorders) | 2 (2)
Infection (Infections and infestations) | 4 (4)
Numbness (Skin and subcutaneous tissue disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | endoAVF (N=100)
Thrombosis (Vascular disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
The study was discontinued prior completion due to company acquisition. Therefore, the full analysis was completed at the 6-month time point for all remaining participants.

Data collection and data management was completed by a third party contractor independent of the sponsor. Statistical analysis was completed per protocol by an independent statistician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT02682420/Prot_SAP_000.pdf